CLINICAL TRIAL: NCT01298349
Title: Perception Processing in Schizophrenia Patients and Normal Population.
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Other Study IDs: 104-10
Record Dates: First submitted 2010-12-02; First posted 2011-02-17 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Schizophrenia; Normal Population
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- schizophrenic patients
- normal population

SUMMARY:
The present study aimed to examine face and object perception processes in schizophrenic patients. Schizophrenia is associated with deficits in visual processing that represent a key feature in the disorder. Previous studies have shown that schizophrenics exhibit deficits in a variety of facial-processing tasks (e.g., face recognition, recognition of facial expressions), that may severely hinder the patients' interpersonal and social skills. Some investigators have attributed these deficits to impairments in configural processing in schizophrenia. That is, an impairment in the ability to process the spatial relations between the constituent parts of a configuration (e.g., the spacing between the eyes of a given face). To date, studies aimed to investigate this possibility (e.g., Schwartz et al., 2002; Yong-Wook et al., 2008) yielded conflicting results. Additionally, it is not yet clear whether the hypothesized impairment in configural processing is restricted to faces, or whether it is more general in nature and applies to objects as well.

DETAILED DESCRIPTION:
In the present study we investigate the relative contribution of component versus configural properties to face and object perception in schizophrenic and control subjects. To this end, we designed a series of experiments that are based on former work by Kimchi and Palmer (1982), and on my Ph.D. dissertation conducted under the supervision of Prof. Ruth Kimchi at the IIPDM.

Experiment 1 investigates the relative roles of local parts versus global configuration in object perception by applying a technique formalized by Kimchi and Palmer (1982). Participants are presented with hierarchical figures, in which larger figures (e.g., a "global" triangle) are constructed by smaller figures (e.g., "local" squares).

Participants (schizophrenics and controls) perform a similarity-judgment task. In each experimental trial, participants are presented with a triad of stimuli: a standard figure and two comparison figures. Participants are asked to determine which of the two comparison figures is more similar to the standard. Each figure consists of a global square or triangle made of local squares or triangles. In the "same configuration" comparison figure different elements are arranged in the same configuration as the standard figure. In the "same element" comparison figure, the same elements as in the standard figure are used, but are arranged in a different configuration. The number of elements used to construct the standard figure is varied. Previous data with normal perceivers (Kimchi & Palmer, 1982) showed that as the number of elements increased (and their sizes decreased) perceivers tended to base their similarity judgments on the global configuration, rather than on its local elements. If schizophrenics are impaired in their ability to process configural information then their similarity judgments should mainly rely on the local elements rather than on the global configuration.

Experiment 2 examines the relative contribution of facial components (e.g., eyes, nose, mouth) versus configural properties (e.g., spacing between the eyes) to face perception, by applying Garner's speeded classification paradigm (Garner, 1974). We have previously applied this paradigm in my Ph.D. dissertation to study face perception in normal perceivers.

The stimulus set consists of four faces created by orthogonally combining components (eyes, nose, and mouth) and configural information (inter-eyes distance and nose-mouth distance). On each trial participants are asked to classify a face on either its components or its configural information, in two conditions. In the control condition only one facial dimension varies (e.g., components) while the other dimension (e.g., configural information) is held constant. In the filtering condition the two dimensions are varied orthogonally. Equal performance in the control and filtering conditions indicates that participants are able to selectively attend to the relevant dimension - the dimensions are processed independently. Poorer performance in the filtering condition than in the control condition - Garner interference - indicates that it is not possible to selectively attend to one dimension while ignoring another, irrelevant dimension - the dimensions are processed interactively.

Results with normal perceivers revealed a symmetric Garner interference with upright faces: participants were unable to selectively attend to components and ignore irrelevant variation in configural information, and vice versa. These results imply perceptual interdependence in processing components and configural information. If schizophrenics are impaired in their ability to process configural information then patients should be able to selectively attend to components and ignore irrelevant variation in configural information, but not vice versa. This pattern would indicate the relative dominance of components over configural properties in upright face processing of schizophrenia patients.

ELIGIBILITY:
Inclusion Criteria:

* schizophrenia or schizo-affective disorder
* normal population with no psychiatric history
* Stable medication for at least a month before participating in the study
* subjects must have normal vision or revised

Exclusion Criteria:

* deterioration of the disorder
* subject will

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients diagnosed with schizophrenia or schizo-affective disorder according to DSM4 and normal population with no psychiatric history
Sampling Method: Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Performance in Experiment 1: Probability of Global Perception (%) | 2 weeks.
  The probabilities (in percentage) of choosing the comparison figure having the same configuration as the standard figure. That is, the ratio between the number of trials in which participants chose the comparison figure as having the same configuration as the standard figure, and the total number of trials.
Performance in Experiment 2: Response Time (milliseconds) | 2 weeks.
  Response Time in milliseconds; will be measured from stimulus onset on screen until prticipant's response.
Performance in Experiment 2: Error Rate (%) | 2 weeks.
  Percentage of Errors; The ratio between number of errors and the total number of responses.

CONTACTS AND LOCATIONS:
Overall Officials: Boaz Bloch, MD, Principal Investigator — Haemek Mediacl Center; Alon Reshef, MD, Study Chair — haemek medical center; Rama Amishav, Phd, Study Chair — haemek medical center
Locations (1):
- Haemek Medical Center, Afula, Israel